CLINICAL TRIAL: NCT04818216
Title: NIRVANA: NIcotinamide Riboside in SARS-CoV-2 pAtients for reNAl Protection
Brief Title: Nicotinamide Riboside in SARS-CoV-2 (COVID-19) Patients for Renal Protection
Acronym: NIRVANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kumar Sharma, Holder of the L. David Hillis, M.D. Endowed Chair, Medicine -Renal Diseases, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20200914H; 3UH3DK114920-04S2 (NIH)
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV-2 Infection; Acute Kidney Injury
MeSH Terms: conditions — COVID-19; Acute Kidney Injury | interventions — microcrystalline cellulose; nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, placebo-controlled clinical interventional trial
Who Masked: Participant, Investigator
Masking Description: The study drug (NR or placebo) packaging and labeling will be designed to maintain the blinding of the investigator's team and the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo capsules will be administered 2 capsules twice daily for 10 days
  Interventions: Drug: Placebo
- Nicotinamide Riboside Group (Experimental): Nicotinamide riboside 250mg capsules will be administered 2 capsules twice daily for 10 days
  Interventions: Drug: Nicotinamide riboside

INTERVENTIONS:
Drug: Placebo — Placebo capsule containing inert ingredient
  Other Names: Microcrystalline cellulose
  Arms: Placebo Group
Drug: Nicotinamide riboside — 250 mg Nicotinamide riboside capsules
  Other Names: Niagen
  Arms: Nicotinamide Riboside Group

SUMMARY:
An interventional clinical trial using oral nicotinamide riboside (NR) in hospitalized patients with COVID-19 infection and acute kidney injury to determine the effect of NR on whole blood nicotinamide adenine dinucleotide (NAD+) levels and to evaluate safety of the use of NR.

DETAILED DESCRIPTION:
The study team chose a treatment protocol with NR as a treatment for patients who will be admitted with COVID-19 related illness and develop AKI after admission. Treatment duration will be for 10 days and the primary study endpoint will be the change in whole blood NAD+ from baseline to end of treatment in NR group vs placebo group. The study team will evaluate whole blood NAD+ levels as a marker of efficacy and biological effect of NR.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form from a participant or legally authorized representative (LAR);
2. Male or female, >18 years old;
3. Hospitalized participants with a laboratory diagnosis of COVID-19 infection
4. Evidence of persistent AKI as defined by the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines (Table 3);
5. Willing to adhere to the study intervention regimen;

Exclusion Criteria:

1. Hypersensitivity to nicotinamide riboside (NR);
2. Pregnant or lactating women confirmed with positive laboratory pregnancy tests as per local requirements;
3. eGFR <15 mL/min/1.73 m2 as per the Chronic Kidney Disease Epidemiology Collaboration equation at admission lab;
4. Maintenance renal replacement therapy or initiation of renal replacement therapy before randomization
5. Currently on NR or nicotinamide or vitamin B3 (niacin) supplementation (multivitamins are allowed);
6. Concomitant cirrhosis of liver or acute liver failure;
7. Any medical history or condition that might, in the opinion of the attending physician, put the participant at significant risk if he/she were to participate in the trial;
8. Individuals with kidney transplant;
9. Individuals with blood platelet count <100,000/microL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Sharma, MD, Principal Investigator — UT Health San Antonio
Locations (4):
- United States (4):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University Health Systems, San Antonio, Texas
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the time when summary data are published or otherwise made available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Started | 13 | 15
Completed | 9 | 13
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Nicotinamide Riboside Group | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.31 (8.25) | 52.40 (15.99) | 52.36 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 6 | 13 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Whole Blood NAD+ Level
Description: Measure of NAD+ level in whole blood from treatment beginning to end
Time Frame: Baseline to 10 days
Population: Analysis set is a modified intention to treat with participants receiving at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Number analyzed (Participants) | 13 | 15
μg/mL | -0.02 (0.02) | 0.06 (.07)

2. Primary Outcome: Number of Participants With Adverse Events of Grade 3 or Higher
Description: Safety of NR in hospitalized patients with COVID-19 and AKI (defined as adverse event of Grade 3 or higher). Not every grade 3 event was considered to be serious.
Time Frame: Baseline to 10 days
Population: Analysis set is a modified intention to treat with participants receiving at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Number analyzed (Participants) | 13 | 15
participants | 8 | 12

3. Primary Outcome: Occurrence of Thrombocytopenia
Description: Number occurrences of thrombocytopenia defined as >25% decline in blood platelet count from baseline.
Time Frame: Baseline to 10 days
Population: Analysis set is a modified intention to treat with participants receiving at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Number analyzed (Participants) | 13 | 15
participants | 1 | 1

4. Secondary Outcome: Change in Area Under the Curve (AUC)
Description: To determine the effect of NR on changes in AUC serum creatinine from baseline during the 10-day intervention
Time Frame: Baseline to 10 days
Population: Analysis set is a modified intention to treat with participants receiving at least 1 dose of study drug.
Measure: Median (Inter-Quartile Range); unit: mg/dL x day
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Number analyzed (Participants) | 13 | 15
mg/dL x day | 17.1 [9.3 to 21.4] | 17.9 [14.9 to 22.8]

5. Secondary Outcome: Effect of NR on Major Adverse Kidney Events (MAKE)
Description: Number of occurrences of MAKE defined as doubling of serum creatinine, the initiation of long-term dialysis, or death from any cause.
Time Frame: 30 days to 90 days
Population: Analysis set is a modified intention to treat with participants receiving at least 1 dose of study drug.
Measure: Number; unit: Number of MAKE events
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Number analyzed (Participants) | 13 | 15
Number of MAKE events | 6 | 12

6. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Description: Measurement of change in eGFR at 30-90 days post randomization
Time Frame: 30 days to 90 days
Population: Analysis set is a modified intention to treat with participants receiving at least 1 dose of study drug. Limited number of participants (n <5) for whom serum creatinine values (change in estimated Glomerular Filtration Rate or eGFR) were available at 30d and 90d.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Number analyzed (Participants) | 3 | 4
mL/min/1.73m^2
  30-day: number analyzed (Participants) | 2 | 4
  30-day | 86.38 (23.35) | 79.02 (58.12)
  90-day: number analyzed (Participants) | 1 | 1
  90-day | 112.08 | 129.91

7. Secondary Outcome: Change in Proteinuria
Description: Measurement of change in proteinuria at 30-90 days post randomization
Time Frame: 30 days to 90 days
Population: Analysis set is a modified intention to treat with participants receiving at least 1 dose of study drug. Proteinuria was not routinely assessed in a hospital setting for COVID patients and an additional measurement was not performed due to infectious concerns.
Arm/Group | Placebo Group | Nicotinamide Riboside Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected with start dates occurring any time after informed consent is obtained until Day 90 - the last visit of the study.
Description: Adverse event severity was graded as per the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Adverse events with Grade 3, Grade 4, and Grade 5 were captured in this trial.
Arm/Group | Placebo Group | Nicotinamide Riboside Group
All-Cause Mortality (participants affected / at risk) | 6/13 | 11/15
Serious Adverse Events (participants affected / at risk) | 7/13 | 12/15
Other Adverse Events (participants affected / at risk) | 6/13 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=13) | Nicotinamide Riboside Group (N=15)
Worsening of renal function requiring dialysis (Renal and urinary disorders) | 3 (3) | 4 (4)
Acute encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute-subacute infarcts in right frontal right parasagittal and right occipital regions (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Septic shock (General disorders) | 1 (1) | 0 (0)
Cardiopulmonary arrest secondary to COVID-19 (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 11 (11) — Includes cause of death non specified in medical records and death due to: COVID-19 Pneumonia Acute respiratory failure with hypoxia Multi-organ system failure Anoxic brain injury secondary to COVID
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=13) | Nicotinamide Riboside Group (N=15)
Elevated liver enzymes (Hepatobiliary disorders) | 0 (0) | 4 (4)
Elevated biliruin (Hepatobiliary disorders) | 0 (0) | 1 (1)
Leukocytosis (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Superficial venous thrombosis of the mid right cephalic vein (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Occlusive deep venous thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Delirium (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT04818216/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04818216/ICF_000.pdf